CLINICAL TRIAL: NCT03510039
Title: Pilot Study Describing the Effect of an Early Nursing Intervention Device on the Anxious Experience of "Third-party" People Who Participate in the First Involuntary Commitment Hospitalization From a Relative
Brief Title: Early Intervention AND NURSING Support for an " Involuntary Commitment Procedure " for a Close Relative
Acronym: Vécu/Tiers/Psy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC31/17/0322; 2017-A03043-50 (Other: ID-RCB)
Record Dates: First submitted 2018-03-09; First posted 2018-04-27 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Anxiety
Keywords: Involuntary commitment hospitalization; close relative
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Mono-centric pilot comparative study like " Before /After ". It will be necessary to recruit at first 35 thirds benefiting from the in current load, "Before" phase, then to set up our intervention, and recruit another 35 different thirds for the "After".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Before" Group (Active Comparator): 35 Thirds benefiting from the usual care
  Interventions: Other: Usual care
- "After" Group (Experimental): Recruit 35 Thirds for the phase phase "After" : Early device / Follow up by nurses
  Interventions: Behavioral: Early device / Follow up

INTERVENTIONS:
Behavioral: Early device / Follow up — Early device:
  Standardized Nursing Interview (30 minutes) with the Third Party Person Measure and follow the anxiety of the Third Party by rating the AMDP-AT scale, on D0 and D7
  Telephone follow-up by nurses:
  Interviews built and standardized, to M2, M4 and M6 Quantification of the AMDP-AT anxiety scale on each call
  Arms: "After" Group
Other: Usual care — Group "Before" : usual care by nurses
  Arms: "Before" Group

SUMMARY:
In a context of first hospitalization under the constraint of a relative in psychiatric emergencies:

* effect of an early intervention and a 6-month nursing follow-up on the anxious experience of third party persons
* effect of nursing support on family dynamics, on the durability of outpatient care and adherence

DETAILED DESCRIPTION:
The patient that is meeting during time travel at Psychiatric Emergency come with their families wich live (or have been lived) the crisis at home, in the street, with their family doctor. With a psychic incoming sufferance, when the patient refuses his medicines, doctors ask to someone close to the patient to become his Third party, his first guarantor of the without consent care commitment. These without consent hospitalizations at Toulouse University Hospital, and all over France hospitals, rise continuously. Our daily nursing exercise is to support those helping people. The sentiment felt by our nursing team during the exchange, underlines ambivalence and several emotional problems and difficulties, which are even harder for a first time occurence.

Patient's close relatives that become a " resource " during non-consensual hospitalization could be affected indirectly by the burden of this referent role. Between culpability, isolation and exhaustion, the studies show that their ability to " resist " is a real help for patient progression. This statement is showed by nursing team (even belonging to others structures) listened during our exploratory investigation.In our professional practice, our specific emergency environment is firstly focused about patient in crisis situation and about his security. In this environment, there is no formerly dedicated time for relatives needing, once actors and public in this acute disease. Relatives hard experiences in a very central moment that we could consider as care beginnings, should impact therapy and patient health care plan. An early, well defined nursing act, built on close relatives needs and expectations could enhance this particular moment that should facilitate the following of the patient disease. A lot of data cited in literature specify the central role of relatives for a psychic patient, but there is no study about an early nursing intervention for Relatives during a psychiatric emergency.

ELIGIBILITY:
Inclusion Criteria:

* Being the "Third Party" adult, during the first involuntary commitment procedure of a close relative, in an ASPDT(u) form.
* Being physically present during the admission, within 24 hours after the arrival of the patient.
* Accept to be recontacted by phone to J7, M2, M4 and M6
* Affiliated person or beneficiary of a social security scheme.
* Free and informed consent, signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research).

Exclusion Criteria:

* To be the guardian or any person in charge of legal representation with the patient.
* Pregnant or lactating woman (the duration of the study may affect the subject's compliance and availability).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-09-13 (Actual)

PRIMARY OUTCOMES:
Effect of early nursing intervention in the short term on the experience of the close relative | 6 month
  Effect of early nursing intervention in the short term on the experience of the close relative compared to current support Measured by the evolution between D0 and D7 (first follow-up call telephone) with the AMDP-AT anxiety scale The AMDP system is a clinical measure of psychopathology. The Association de Methodology and Documentation in Psychiatry has developed this system of standardized quantification of psychopathology This is a synthetic version of 17 anxiety items (with a score included between 0 and 68), which is therefore a shorter scale than the full AMDP scale The AMDP-AT is particularly adapted to our emergency situation to assess the experience of the close relative, because it takes into account the multiple dimensions at the moment of the immediate anxiety situation

SECONDARY OUTCOMES:
Number of visits to the attending physician, consultations at the Psychological health center | 6 months
  Number of visits to the attending physician, consultations at the Psychological health center, appeals psychiatric emergencies, psychiatric emergency room visits and hospital admissions possible, patients whose close relative has benefited from the "After" phase, compared to in current load, counted by calls for both groups to M2, M4 and M6. The calls will be non-interventional for the "Before" phase, and formalized interventional for the phase "After"
Effect of nurse intervention over the medium term on the experience of the close relative | 6 months
  Effect of the intervention of the nurses in the medium term on the experience of the close relative, measured by the change between J0 and M6 by Telephone Tracking Calls with Anxiety Scale AMDP-AT

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre CASTANET, nurse, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No